CLINICAL TRIAL: NCT02712632
Title: Genetics of Diabetes Audit and Research in Tayside and Scotland
Acronym: GoDARTS
Status: Completed | Type: Observational
Sponsor: University of Dundee (Other)
Responsible Party: Sponsor
Other Study IDs: 2016DM03 GoDARTS-Scotland
Record Dates: First submitted 2016-02-12; First posted 2016-03-18 (Estimated); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At visit 1 blood samples will be collected for DNA and RNA extraction. Urine samples will be collected to measure for biomarkers. Stool samples will be collected to measure for microbiota. (Stool samples will only be collected from those patients who are initiated on metformin therapy during the study period.
  For those patients who are commenced on metformin therapy during the study a second study visit is required where all blood, urine and stool samples will be repeated.
Oversight: Data Monitoring Committee: No

SUMMARY:
The GoDARTS study will encompass all patients, with diabetes, aged 16 and upwards who meet the planned inclusion criteria. The study aims to investigate biomarkers associated with diabetes progression, therapeutic response, diabetes complications and related traits, and specifically to investigate mechanisms of action and response to metformin. The study will specifically target patients who have been diagnosed within the past 2 years and follow up will be by linkage to electronic health record data. Up to 6,000 patients will be recruited into the study over a period of 2-3 years with a primary aim to identify 1000 of these patients who should be suitable to be started on metformin therapy.

Most patients will undergo a single screening visit lasting approximately 20 minutes conducted on an outpatient basis. Patients commenced on metformin therapy will need to attend a second clinic visit to be carried out between 4-6 months after initiation of metformin therapy.

Up to 9 health boards will be approached regarding participating in the study, and it is estimated that between 4-6 diabetes patients will be recruited into the study each week, at each site.

All screened patients will provide consent for data linkage and longitudinal follow up and their samples and data will be used to supplement the SHARE/SDRN bioresource. The collection into the resource will be managed by the co-ordinating centre study team based at the University of Dundee/NHS Tayside. The resource will be hosted by the Tayside Biorepository and access to samples and data will be managed by the Tayside Biorepository on behalf of the whole of Scotland.

DETAILED DESCRIPTION:
This GoDARTS-Scotland proposal aims to investigate biomarkers associated with diabetes progression, therapeutic response, diabetes complications and related traits, and specifically to investigate mechanisms of action and response to metformin. GoDARTS-Scotland will specifically target the patient group who have been diagnosed with diabetes in the previous 2 years and follow up will be by linkage to electronic health record data.

The study will, for the most part, involve a single study visit lasting approximately 20 minutes. Informed consent will be obtained before any study procedures are carried out.

In addition, those patients who are not on metformin will undergo more comprehensive sampling and a second visit, between four to six months, after initiation of metformin. As current guidelines suggest all patients who are newly diagnosed with type 2 diabetes should be treated with metformin the investigator will ask the patient and General Practitioner to consider initiation of metformin, although this is a clinical decision that will be made by the GP. Between four to six months after commencement of Metformin the patient will be asked to return to the clinic for a second visit where additional samples and measures will be taken.

The investigator plans to recruit patients aged 16 and upwards with a diagnosis of diabetes from several Scottish Health Boards.

The Resource will be hosted by the Tayside Biorepository which is part of the East of Scotland Tissue Bank. Access to samples and data will be managed by the Tayside Biorepository on behalf of the whole of Scotland. All initial requests for access will be made to the Tayside Biorepository Access Committee who will manage the process and send requests for access to data to the relevant access committees.

All eligible patients will be recruited into this study from February 2016 until January 2019 and this will allow any necessary follow up visits to take place.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 16 and over.
* Diagnosis of diabetes within the past 2 years.
* Either Non-Type 1 diabetes controlled by diet only with an HbA1c ≥ 48; or Type 1 diabetes
* Able to give informed consent.

Exclusion Criteria:

* Patients with non-type 1 diabetes who have had previous treatment with insulin or an OHA or GLP-1.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients for this study will be identified from the SDRN and SHARE Research Registers. (These patients have given prior consent to be contacted about research studies.)
  Patients will also be selected from secondary and primary care clinics.
Sampling Method: Probability Sample
Enrollment: 1227 (Actual)
Dates: Start 2016-06-20 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
HbA1c reduction. | 6 months to 1 year
  For the primary analysis on the determinants of metformin response the primary outcome is HbA1c reduction

CONTACTS AND LOCATIONS:
Overall Officials: Ewan Pearson, MBBChir PhD, Principal Investigator — University of Dundee and NHS Tayside
Locations (1):
- University of Dundee, Dundee, Tayside, United Kingdom